CLINICAL TRIAL: NCT04462289
Title: Electronic Proactive Outreach for Smokers With COPD: Engaging Patients to Quit (CDA 19-081)
Brief Title: Electronic Proactive Outreach for Smokers With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDX 20-001
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Smoking
Keywords: smoking cessation; Pulmonary Disease, Chronic Obstructive; implementation science
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Patient-level randomized pilot
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Randomly assigned sample who will receive usual care for tobacco cessation treatment
- Proactive Outreach (Experimental): Randomly assigned sample who will receive a proactive offer of tobacco treatment with connection to motivational texting program.
  Interventions: Behavioral: Proactive Outreach

INTERVENTIONS:
Behavioral: Proactive Outreach — Motivational electronic offer of tobacco cessation support via motivational texting program with care connection to patient's choice of smoking cessation programs
  Arms: Proactive Outreach

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common respiratory diseases, with 90% of cases directly attributable to smoking. Unfortunately, many patients continue to smoke and have an urgent need to quit. Proactive tobacco treatment programs identify patients outside of a routine clinical appointment and engage them in making a supported quit attempt.

Most previous research of proactive tobacco treatment has used telephone outreach, which can be resource intensive. Electronic methods (texting, secure messaging) may be effective while requiring fewer resources.

In this study, the investigators will adapt a clinically available motivational texting program with content tailored to smokers with COPD. First, information will be gathered from smokers with COPD and the medical staff who care for them to adapt the program for electronic delivery. Then, the program will be pilot-tested. Smokers with COPD will be randomly assigned to either usual medical care or the outreach intervention, with goals to increase participation in smoking cessation programs, quit attempts, and successful cessation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the most common respiratory conditions and the 4th leading cause of death in the US. 90% of cases are directly attributable to smoking. Quitting smoking is the most important intervention for these patients, who continue to smoke at rates double the national average. Smokers with COPD remain undertreated for tobacco use. Proactive tobacco treatment programs identify patients outside of a routine clinic visit, engage them in making a quit attempt and connect them with treatment. These programs may be particularly beneficial for smokers with COPD. Previous phone-based programs are resource intensive to deliver. Electronic methods for delivering proactive outreach for tobacco cessation may be effective and cost-effective, and can be tailored to the target population.

Hypothesis: A proactive tobacco treatment program delivered electronically and tailored to smokers with COPD will be effective and cost effective for increasing quit engagement among smokers with COPD.

Study design: Multi-aim implementation study with randomized pilot. Aim 1: Mixed methods (survey and interview) assessment of current use of health information technology among smokers with COPD with a focus on the impact of the chronic disease state on tobacco cessation.

Aim 2: Qualitative assessment of barriers and facilitators to implementation of proactive tobacco treatment programs for patients with COPD among staff and leadership.

Aim 3: Randomized pilot of a proactive tobacco treatment program for smokers with COPD delivered through text messaging.

ELIGIBILITY:
Inclusion Criteria:

* Veterans active in clinical care (at least one primary care or pulmonary visit within the past year)
* Past-year smoking status in the electronic health record indicating current smoking, confirmed on enrollment call
* Diagnosed with COPD (2 International Classification of Diseases (ICD)-10 diagnoses of COPD within the past 2 years)
* Currently enrolled in MyHealtheVet secure messaging

Exclusion Criteria:

* Already enrolled in behavioral VA tobacco treatment
* Enrolled in hospice
* Undergoing active cancer treatment
* Advanced dementia
* Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne C. Melzer, MD MS, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were identified using the electronic health record (EHR) with: 2 or more ICD-10 codes for COPD in the past 2 years at any VA healthcare system, along with a visit to primary care or pulmonary medicine at the Minneapolis VA Health Care System with in the past 18 months, and their last tobacco assessment indicated current smoking. Participants were excluded if they were enrolled in hospice, a malignancy, had advanced dementia, enrolled in a tobacco treatment program.
Period: Overall Study
Arm/Group | Usual Care | Proactive Outreach
Started | 41 | 83
Completed | 36 | 72
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 4 | 5
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Proactive Outreach | Total
Number analyzed (Participants) | 41 | 83 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.93) | 68.9 (7.22) | 68.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 35 | 68 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 75 | 114
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 3 | 8 | 11
  White | 33 | 64 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 8 | 9
Rurality [Count of Participants; unit: Participants]
  Highly Rural | 1 | 0 | 1
  Rural | 18 | 37 | 55
  Urban | 22 | 46 | 68
  Missing | 0 | 0 | 0
Education Attainment [Count of Participants; unit: Participants]
  Less than High School | 2 | 3 | 5
  High School Granduate/GED | 15 | 23 | 38
  Some College or Vocational Education | 19 | 38 | 57
  College Graduate/Post-Graduate | 5 | 19 | 24
Cigarettes per Day [Count of Participants; unit: Participants]
  10 or fewer | 16 | 26 | 42
  11 to 20 | 20 | 47 | 67
  21 or more | 5 | 10 | 15
Past Year Quit Attempts [Count of Participants; unit: Participants] | 27 | 36 | 63
No particular timeframe to Quit [Count of Participants; unit: Participants] | 20 | 54 | 74
Heaviness of Smoking Index [Mean (Standard Deviation); unit: units on a scale] — This is a calculated scale that measures nicotine dependence using two questions: how soon after waking do you smoke your first cigarette and cigarettes per day. Scores range from 0-6. Lower numbers correspond with lower nicotine dependence.
  Question 1: Time to First Cigarette After waking:
  6-30 min: 3 pts 31-60 min: 2 pt after 60 min: 0 pt
  Question 2: Cigarettes per day 10 or fewer: 0 pt 11-20: 1 pt 21-30: 2pt 31+ : 3pt
  calculated by adding points from each question
  Dependence level:
  low: 0-2 pt medium: 3-4 pts High: 5-6 pts
  units on a scale | 2.41 (1.61) | 2.48 (1.42) | 2.46 (1.48)
Quit Ladder [Count of Participants; unit: Participants]
  I don't want to stop/I should stop smoking but don't really want to | 14 | 25 | 39
  I want to stop smoking but haven't thought about when | 4 | 13 | 17
  I really want to stop smoking, but I don't know when I will | 6 | 16 | 22
  I want to stop smoking and hope to soon | 2 | 12 | 14
  I really want to stop smoking and intend to in the next 1 or 3 months | 15 | 17 | 32
Use of Texting Every Day [Count of Participants; unit: Participants] | 33 | 64 | 97

OUTCOME MEASURES:

1. Primary Outcome: Participation in Tobacco Cessation Treatment
Description: Any participation in tobacco cessation treatment (medication use, counseling)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 9 | 29

2. Secondary Outcome: 30-Day Abstinence
Description: Number of participants who had not smoked any cigarettes in the past 30 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 2 | 6

3. Secondary Outcome: Quit or Cut Down
Description: Number of participants who have either not smoked in the past 7 days or have cut down in heaviness or frequency
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 12 | 32

4. Secondary Outcome: 7-day Abstinence
Description: Count of participants who have not smoked in the past 7 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 3 | 8

5. Secondary Outcome: Moved Upward on the Quit Ladder
Description: Count of participants who indicated that they were more interested in quitting smoking than at baseline
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 13 | 23

6. Secondary Outcome: Cut Down in Heaviness of Smoking
Description: Cut down by 10 cigarettes per day or in frequency of smoking from daily to some days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 9 | 25

7. Secondary Outcome: Care Coordination
Description: Proportion of participants who completed a care coordination call
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 1 | 11

8. Secondary Outcome: Number of Quit Attempts
Description: Self-reported attempts to quit smoking
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants | 21 | 35

9. Secondary Outcome: Types of Assistance Used
Description: count of the types of assistance participants used
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants
  Medications Alone | 8 | 20
  Medications and Cessation Clinic or Group Class | 0 | 4
  Cessation Clinic or Texting/App Alone | 4 | 1
  Did not use tobacco cessation assistance | 29 | 58

10. Secondary Outcome: Medications Used
Description: count of participant split by tobacco treatment medications used during quit attempts
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive Outreach
Number analyzed (Participants) | 41 | 83
Participants
  Single Nicotine Replacement | 4 | 15
  Combination Nicotine Replacement | 3 | 4
  Varenicline | 1 | 2
  Bupropion | 0 | 2
  did not use medication | 33 | 60

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Proactive Outreach
All-Cause Mortality (participants affected / at risk) | 0/41 | 3/83
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/83
Other Adverse Events (participants affected / at risk) | 0/41 | 0/83

LIMITATIONS AND CAVEATS:
This was a small, single center pilot including mostly white, male Veterans. Results may therefore not be generalizable to other settings. However, this is a group expected to be particularly refractory to treatment. We chose to make relatively moderate adaptations to an existing protocol and there may have been other areas that would have benefitted from further tailoring. Outcomes were relatively short and measured by self-report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04462289/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04462289/ICF_000.pdf